CLINICAL TRIAL: NCT06465732
Title: A Randomized Controlled Study to Evaluate the Efficacy and Safety of Dupilumab in Combination With Short-term Low-dose Tofacitinib in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety of Dupilumab in Combination With Tofacitinib in Moderate to Severe Adult AD Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR2024072
Record Dates: First submitted 2024-06-04; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; tofacitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dupilumab plus tofacitinib (Experimental): this arm receives dupilumab injection and oral tofacitinib.
  Interventions: Drug: Dupilumab; Drug: Tofacitinib
- dupilumab mono (Active Comparator): this arm receives dupilumab treatment only.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — the active comparator arm receive dupilumab only
Drug: Tofacitinib — the experimental arm receive dupilumab plus tofacitinib.
  Arms: dupilumab plus tofacitinib

SUMMARY:
Atopic dermatitis (AD) is a common chronic inflammatory skin disease characterized by intense pruritus and sleep disturbances. The clinical manifestations of AD are varied, with the most basic features being dry skin, chronic eczema-like dermatitis, and intense pruritus. The prevalence in children and adults is about 30% and 10%, respectively. Most patients respond well to topical anti-inflammatory drugs, but approximately 10 percent of patients with moderate-to-severe AD require one or more systemic therapies to achieve good disease control. Although nonspecific immunosuppressive drugs (including glucocorticoids, cyclosporine A, methotrexate, azathioprine, or mycophenolate mofetil) are effective in alleviating or controlling these disorders to some extent, their overall efficacy in patients is limited and associated with significant side effects with long-term use.

The main hallmarks of systemic type II inflammation are eosinophilia and elevated serum immunoglobulin E (IgE) levels. Type II inflammatory response is not only associated with allergic reactions, but is also a driver of such diseases. The release of cytokines (interleukins 4, 5, and 13) in the response to type II inflammation can trigger a lymphocyte-mediated type II inflammatory response, inducing the onset and progression of allergic diseases. Reducing the inflammatory response by inhibiting the above-mentioned inflammatory factors is a potential therapeutic means for the treatment of allergic diseases represented by AD.

Investigational drug Dupilumab injection, an interleukin-4 receptor α (IL-4Rα) antagonist, is a human monoclonal antibody that binds IL-4Rα and inhibits IL-4 and IL-13 signaling. With a molecular weight of about 147 kDa, it inhibits the signaling of interleukin 4 and interleukin 13 and blocks its signaling pathway through the atopic binding of the interleukin 4Ra subunit shared with the interleukin 4 and interleukin 13 receptor complex, and blocks their signaling pathways, which can achieve continuous, efficient and safe improvement of skin lesions, itching and other symptoms and alleviate the condition.

Tofacitinib is a Janus kinase (JAK) inhibitor. JAK is an intracellular enzyme that conducts signals generated by cytokine or growth factor-receptor interactions on cell membranes, thereby affecting cell hematopoiesis and cellular immune function.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the content of the research and voluntarily sign the ICF.
2. 18 years old≤ age ≤ 60 years old (calculated from the date of signing the ICF), male or female.
3. The diagnosis of AD at screening meets the consensus criteria for dermatology in the United States (2014) (see Appendix), and the disease has been in condition for ≥ half a year before screening, and all of the following conditions are met at screening and randomization:

   A. EASI score ≥ 12 points at screening and randomization; B. IGA score ≥ 3 points at screening and randomization (0-4 points IGA scale, 3 points are moderate, 4 points are severe); C. AD involvement of BSA ≥10% at screening and randomization; D. Weekly average of daily peak pruritus NRS score at randomization ≥ 4 points.
4. Subjects of childbearing potential and their partners agree to use effective contraceptive measures throughout the study period (from signing the ICF to 3 months after the last study drug administration) .
5. Able to communicate well with the investigator and comply with the follow-up requirements of the protocol.

Exclusion Criteria:

Subjects with any of the following cannot be enrolled in this study:

1. Allergy to any ingredient in dupilumab or tofacitinib, or allergy or intolerance to other oral JAK inhibitors.
2. Use of any of the following medications or treatments:

   1. Received treatment with other oral JAK inhibitors within 1 month prior to baseline, or lack of efficacy/intolerance to other oral JAK inhibitors in the past, including but not limited to baricitinib, upadatinib and abuxitinib;
   2. Use of excessive pilumab within 6 weeks prior to baseline;
   3. Within 3 months (or within 5 drug half-lives, whichever is longer) prior to baseline, use of other systemic biologics other than dupilumab that are known or likely to affect AD (such as IL-13 receptor antibody [tracilumab], IL-31Rα antibody [nimolizumab], etc.);
   4. Within 4 weeks (or within 5 half-lives, whichever is longer) prior to baseline, have used any kind of systemic therapy for AD: immunosuppressants (such as cyclosporine, methotrexate, azathioprine, mycophenolate mofetil, etc.), glucocorticoids, PDE-4 inhibitors, etc.;
   5. Treatment with phototherapy (narrowband ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + ultraviolet A [PUVA]), tanning bed, or any other luminescent device within 4 weeks prior to baseline;
   6. Allergen-specific immunotherapy (desensitization therapy) within 6 months prior to baseline;
   7. Vaccination with any live vaccine or live attenuated vaccine within 12 weeks prior to baseline; or anticipated need to receive a live or live attenuated vaccine during the study, including at least 12 weeks after the last dose of the investigational drug;
   8. Treatment with any drug or medical device clinical study within 3 months prior to baseline or within 5 half-lives of the drug (whichever is longer, if known), or currently enrolled in another interventional study.
3. Laboratory abnormalities that meet any of the following criteria during the screening period:

   1. Hemoglobin < 90.0 g/L;
   2. White blood cell count< 2.5×109/L;
   3. Neutrophil count< 1.5×109/L;
   4. Lymphocyte count<0.8×109/L;
   5. Platelet count< 100×109/L;
   6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin (TBIL) >2×ULN;
   7. Serum creatinine> 1.2 times ULN; h Any clinically significant other laboratory test abnormalities (as judged by the investigator) that may interfere with the evaluation of the results of this study.
4. Have a history or abnormality of any of the following:

   1. Presence of other cutaneous comorbidities other than AD that may interfere with study assessments;
   2. Subject has active/severe concomitant disease/symptoms (e.g., unstable chronic asthma, etc.) that may require systemic hormonal therapy or interfere with study participation, or requires active and frequent monitoring;
   3. Have a history of 2 or more episodes of herpes zoster, or have a history of disseminated (even a single episode) of herpes zoster, or disseminated (even a single episode) of herpes simplex infection;
   4. Active tuberculosis or γ-interferon release assay at screening (e.g., QUANTIFERON-TB® GOLD, T-SPOT. TB TEST OR OTHER γ-INTERFERON RELEASE ASSAY EQUIVALENT INDEX) IS POSITIVE
   5. Hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), or syphilis infection:
   6. Active skin infection, non-skin infection, or other persistent/chronic infection or invasive infection, which meets the following conditions: 1) skin infection: including bacterial, fungal or viral infection, requiring systemic treatment within 4 weeks prior to the baseline visit, or superficial skin infection within 1 week prior to the baseline visit, or may affect the evaluation of AD lesions; 2) Non-skin infection: need to be given systemic non-gastrointestinal anti-infective therapy within 4 weeks before the baseline visit, or need to receive oral anti-infective therapy within 2 weeks before the baseline visit; 3) Persistent/chronic infection: such as chronic recurrent infection and/or active viral infection such as chronic pyelonephritis, bronchiectasis or osteomyelitis, which is judged by the investigator to be unsuitable for participating in this study; 4) Invasive infection: known history of invasive infection (e.g., listeriosis and histoplasmosis).
   7. Patients who have had thromboembolism (including deep vein thrombosis, pulmonary embolism, arterial thrombosis, etc.) in the past, or other high-risk groups prone to thromboembolism (such subjects are not suitable for participation in this study as judged by the investigator based on clinical evaluation);
   8. Has any of the following history/abnormalities of cardiovascular disease: 1) moderate to severe congestive heart failure (New York Heart Association Class III or IV); 2) Cerebrovascular accident, myocardial infarction, coronary artery stent implantation; 3) poorly controlled or refractory hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥100 mmHg after drug control); 3) There are significant abnormalities in the ECG examination, and participation in the clinical study may pose unacceptable risks to the subject as judged by the investigator, including but not limited to severe arrhythmias, QT interval (QTcF) corrected for heart rate using Fridericia's formula, >480 ms (see Appendix 10 for the calculation formula); 4) Other cardiovascular-related abnormalities/medical history, which, in the judgment of the investigator, are not suitable for participation in this study.
   9. Has a history of gastrointestinal perforation (except appendicitis or penetrating injury), diverticulitis;
   10. Conditions that may interfere with drug absorption, including, but not limited to, short bowel syndrome, gastrectomy, or specific types of bariatric surgery (e.g., gastric bypass); Subjects with a history of gastric banding/segmentation were not excluded;
   11. Those who have a history of lymphoproliferative disorders, or have relevant symptoms/signs that have not been ruled out of lymphoproliferative disorders;
   12. History of any malignancy, with the exception of successfully treated non-melanoma skin cancer (NMSC) or localized carcinoma in situ of the cervix;
   13. Organ transplant patients, who require continuous use of immunosuppressants;
   14. History of drug or alcohol abuse within 6 months prior to screening;
   15. Have a history of nodules or masses (e.g., pulmonary nodules, thyroid nodules, incomplete resection), malignancy cannot be ruled out or there is a possibility of malignant progression, and close observation is required as assessed by a specialist (at least once every six months);

   p Have undergone major surgery within 8 weeks prior to baseline;

   q Has other clinically significant medical conditions that may affect the subject's participation in this study or make the subject no longer suitable to receive an investigational drug product as a candidate (such as any disease that, in the judgment of the investigator, would put the subject at risk for safety by participating in the study, or any disease during the study that would affect the efficacy or safety analysis if the disease/condition worsens).
5. Pregnant or lactating women, or women who plan to become pregnant or breastfeeding during the study.
6. Any reason that, in the opinion of the investigator, would preclude the subject's participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a ≥75% reduction from baseline in Eczema Area and Severity Index (EASI) score (EASI-75) at 16 weeks | 16 weeks

SECONDARY OUTCOMES:
Percentage of participants with an Investigator Global Scoring Method (IGA) score of 0 or 1 at W16 | 16 weeks
Percentage of participants achieving EASI-75 at W12 | 12 weeks
Percentage of participants with an IGA score of 0 or 1 at W12 | 12 weeks
Percentage of participants achieving EASI-90 at W12 | 12 weeks
Percentage of participants achieving EASI-90 at W16 | 16 weeks
Percentage of participants with a ≥4-point reduction from baseline in the weekly mean of the Daily Peak Pruritus Numeric Assessment Scale (NRS) score at W12 | 12 weeks
Percentage of participants with a ≥4-point reduction from baseline in the weekly mean of the Daily Peak Pruritus NRS score at W16 | 16 weeks
Percentage of atopic dermatitis control tool (ADCT) score less than 7 at W12 | 12 weeks
Percentage of atopic dermatitis control tool (ADCT) score less than 7 at W16 | 16 weeks

IPD SHARING:
Plan to Share IPD: Undecided